CLINICAL TRIAL: NCT03386747
Title: Survive and Thrive in Brazil: Boa Vista Early Childhood Program
Brief Title: Survive and Thrive Boa Vista Early Childhood Program
Acronym: STBV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Collaborators: The University of The West Indies (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Inter-American Development Bank (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Alexandra Brentani, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TTS180818280
Record Dates: First submitted 2017-12-13; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Neonatal Death; Mental Competency
Keywords: child development; neonatal mortality
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Masking Description: Treatment requires active participation and will be revealed immediately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Visiting Group (Experimental): Intervention: Home visits to improve parenting behaviors
  Interventions: Behavioral: Home visits to improve parenting behaviors
- Center based parenting group (Experimental): Intervention: Center based parenting groups
  Interventions: Behavioral: Center based parenting groups
- control group (No Intervention): The rest of pregnant women and their children who will not receive the intervention

INTERVENTIONS:
Behavioral: Home visits to improve parenting behaviors — Caregivers will be visited twice per month starting from the third trimester in pregnancy up to age three to discuss important health and development behaviors.
  Arms: Home Visiting Group
Behavioral: Center based parenting groups — Caregivers will be invited to early childhood development groups. Groups will meet at nearby centers twice per month. Caregivers will be invited to participate starting from the third trimester up to age 3 of the child.
  Arms: Center based parenting group

SUMMARY:
The proposed project will tackle the two most salient problems for children under 5 in Brazil: the continued high rates of neonatal mortality, and the large disparities in early childhood development. We propose to extend and scale up previously tested and validated home visiting programs to the city of Boa Vista in the north region of Brazil. The core intervention of the program will be home visits or group meetings to mothers and caregivers by trained child development agents. At the core of the program is a detailed curriculum, which contains gestation and age-specific topics of child health and development to be discussed with caregivers at each encounter.

DETAILED DESCRIPTION:
Even though much progress has been achieved in child mortality globally, relatively minor improvements have been realized in the first four weeks of children's life generally referred to as the neonatal period. Each year, four million infants die within the first 28 days of their life globally. As pointed out in the Lancet's neonatal survival series, 3 million neonatal deaths could be prevented each year by low-cost interventions. In Brazil, more than 25,000 newborns die each year within the first 28 days of their life, with a majority of deaths occurring in the first week. Previous studies suggest that one of the most effective ways to prevent such deaths are home visiting programs, which support mothers in the first weeks of infant's lives, promote breastfeeding and kangaroo mother care, and ensure appropriate medical care when needed. From a child health and child development perspective, optimal outcomes appear only feasible if continued support is provided to mothers from pregnancy throughout the first years of children's life. Home-based visits and support have become increasingly recognized as a both crucial and highly cost-effective strategy to achieve such outcomes.

The objective of this project is to extend and scale up the previously tested and validated home visiting programs to the city of Boa Vista. At the core of this program is a detailed curriculum, which contains gestation and age-specific topics of child health and development to be discussed with caregivers at each home visit. The intervention package will start in the third trimester of pregnancy and feature to sessions per month up to age 3 years.

This curriculum will be delivered through two separate - and randomly assigned - platforms: home visits through trained Child Development Agents (CDAs), and center-based delivery of the same delivery to groups of caregivers. The pilot study in Sao Paulo suggests that each CDA can handle approximately 40 families, visiting each caregiver twice per month. Visits will be initiated during the second trimester of pregnancy. The visits during pregnancy will not be a substitute for prenatal care but are designed to prepare mothers for babies and set up a relationship for a closer follow-up after birth. In Brazil, as well as globally, the numbers of pre-term deliveries and stillbirth is rather large, 20% of mature stillbirths (more than 37 weeks of gestation, more than 2.5 Kg) so the pre-natal care can be improved clearly. The visits would also occur during the neonatal period, when the largest proportional of under 5 mortality happens. This would be the first component of the program, addressing maternal and perinatal/neonatal mortality. Particular attention will be given to mothers after birth, with two special visits scheduled for the first week after birth focusing on maternal mental health; breastfeeding as well as kangaroo mother care when appropriate. Such visitation programs have been successfully tested within the family health strategy, and will be further reinforced and complemented by the new visitation program.

The city of Boa Vista has a population of approximately 330,000 people, with, 22,377 families (~30%) currently receiving social cash transfers under the bolsa familia program. The city is comparable to the national average in terms of the observed poverty rates, and roughly average in terms of its size. Infant mortality rate is estimated at 14.2 per 1000 live births, with 21% of births given by teenage mothers and 15% of infants born preterm.

The proposed project will exclusively target the most vulnerable households currently supported by the bolsa familia social cash transfer program. According to municipality estimates, about 5000 children are born each year in eligible households.

ELIGIBILITY:
Inclusion Criteria:

- pregnant women living in the urban area of Boa Vista

at LEAST ONE of the following vulnerability criteria

1. bolsa família or other social cash transfer program recipient
2. household income per capita less than half of minimum wage
3. previous exposure to domestic or sexual violence before.

Exclusion Criteria:

* women living outside of Boa Vista urban area
* women not meeting social vulnerability criteria above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall child development - PRIDI score | Age 2 - year 3 of the study
  Children's overall development will be assessed using the PRIDI child development assessment tool.

SECONDARY OUTCOMES:
Neonatal mortality | 3 years
  Probability of death between day 0 and day 27 after birth

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Brentani, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brentani A, Ferrer APS, Bessa L, Chang S, Walker S, Powell C, Hamadani J, Grisi S, Fink G. Survive and Thrive in Brazil: The Boa Vista Early Childhood Program: study protocol of a stepped-wedge, randomized controlled trial. Trials. 2020 May 7;21(1):390. doi: 10.1186/s13063-020-4217-3. PMID 32381097